CLINICAL TRIAL: NCT03791476
Title: A Phase I/II,Single Center,Randomized,Double-Blind,Placebo-Controlled Study to Evaluate the Feasibility of Using Human Recombinant C1 Inhibitor(RUCONEST®) as a Therapeutic Strategy to Reduce the Incidence of Delayed Graft Function in Recipients of Kidneys From Donation After Cardio-Circulatory Death
Brief Title: RUCONEST® as a Therapeutic Strategy to Reduce the Incidence of Delayed Graft Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-1325; A539742 (Other: UW Madison); SMPH/SURGERY/TRANSPLANT (Other: UW Madison); Protocol Version 12/26/2019 (Other: UW Madison)
Record Dates: First submitted 2018-07-12; First posted 2019-01-02 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-07

CONDITIONS: Kidney Failure
Keywords: Delayed graft function
MeSH Terms: conditions — Renal Insufficiency; Delayed Graft Function | interventions — conestat alfa; Saline Solution

STUDY DESIGN:
Intervention Model Description: Intervention versus placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Intervention is saline solution placebo (0.9% Sodium Chloride IV to equal volume of investigational arm: intraoperatively, and then every 12 hours x 2 = total of 3 doses)
  Interventions: Other: Saline Solution
- rhC1INH (Experimental): Intervention is rhC1INH 100 U/kg intraoperative followed by 50 U/kg every 12 hours x 2 = total of 3 doses (200 U/kg)
  Interventions: Drug: rhC1INH

INTERVENTIONS:
Drug: rhC1INH — C1 esterase inhibitor
  Other Names: ruconest
  Arms: rhC1INH
Other: Saline Solution — saline solution
  Arms: Control Group

SUMMARY:
An unmet medical need exists for therapeutic regimens in transplantation that allow immediate postoperative graft function, thereby improving graft survival. Delayed graft function (DGF) after transplantation is the most common complication affecting kidney allographs in the immediate transplant period. The specific aim of this study is to evaluate the effect of recombinant human C1-inhibitor (rhC1INH), as a kidney recipient intra- and post operative treatment strategy to decrease systemic inflammation and decrease the incidence of DGF from donation after cardiac death donors (DCD).

DETAILED DESCRIPTION:
This is a randomized, single-center double blinded study.

The main objective of this study are to determine the ability of rhC1INH to reduce the incidence and severity of delayed graft function in comparison to placebo in recipients of kidneys after cardio-circulatory determination of death (DCD).

This trial has specifically been designed to evaluate the protective effect of rhC1INH treatment in patients at high risk of developing DGF. The selection of potential donors to be part of this study will be limited to the population of DCD donors which have historically shown a risk of developing DGF ranging between 40-55%. Participation in each group will be randomly assigned. Treatment will be administered by an intra-operative infusion of placebo or rhC1INH (100 Units/kg) IV followed by twice a day infusion of 50 Units/Kg IV for the following 48 hours.

A total of 20 subjects will be divided into 2 groups:

Group 1: Control group: standard recipient management + placebo (0.9% Sodium Chloride IV to equal volume of investigational arm: intraoperatively, and then every 12 hours x 2 = total of 3 doses). treatment (n=10) Group 2: Standard recipient management + 100 U/kg intraoperative followed by 50 U/kg every 12 hours x 2 = total of 3 doses (200 U/kg).

Max dose 8400 units for the initial dose and 4200 units maximum for the second and third doses.

ELIGIBILITY:
Inclusion Criteria for Transplant Recipient:

Adult patients receiving a transplanted kidney should satisfy the following to be considered part of the study:

1. Has the ability to understand the requirements of the study, is able to provide written informed consent (including consent for the use and disclosure of research related health information).
2. Male or female at least 18 years of age.
3. Is to be a recipient of a transplant from a deceased donor (donation after cardio-circulatory determination of death criteria).
4. Is able to comply with standard of care induction therapy requirement, such as antibody induction therapy with rabbit polyclonal anti-thymocyte globulin,anti-CD25 (anti-IL2R), or Anti-CD52.
5. A female subject is eligible to enter the study if she is:

   1. Not pregnant or nursing
   2. Of non-childbearing potential (i.e., post-menopausal defined as having been amenorrheic for at least 1 year prior to screening, or has had a bilateral tubal ligation at least 6 months prior to administration of study drug or bilateral oophorectomy or complete hysterectomy).
   3. If of childbearing potential, must have a negative serum pregnancy test within 48 hours prior to transplant surgery and be using an effective means of contraception (per the site-specific guidelines or using 2 methods of birth control concurrently, whichever is more stringent) which will be continued until the Day 180 visit.
6. Male subjects with female partners of childbearing potential must agree to use an effective means of contraception (per the site-specific guidelines or use 2 methods of birth control concurrently, whichever is more stringent), which will be continued until the Day 180 visit. They will also agree not to donate sperm until 6 months after dosing.
7. Must be up-to-date on cancer screening according to site-specific guidelines and past medical history must be negative for biopsy-confirmed malignancy within 5 years of randomization, with the exception of adequately treated basal cell or squamous cell carcinoma in situ or carcinoma of the cervix in situ.
8. Must be willing to comply with the protocol procedures for the duration of the study, including scheduled follow-up visits and examinations.

Exclusion Criteria for Transplant Recipients:

1. Use of an investigational drug in the 30 days before surgery.
2. Participation in any other research study (drug or non-drug) without prior approval from the sponsor investigator.
3. Recipient of a live donor kidney or a kidney from a brain death donor (DBD) donor.
4. Recipient of donor kidney preserved with normothermic machine perfusion.
5. Scheduled to undergo multiorgan transplantation.
6. Has a planned transplant of kidneys that are implanted en-bloc (dual kidney transplantation).
7. Has planned transplant of dual kidneys (from the same donor) transplanted not en-bloc.
8. Has lost first kidney transplant due to graft thrombosis.
9. Is scheduled for transplantation of a kidney from a donor who is known to have received an investigational therapy under another IND/CTA for ischemic/reperfusion injury immediately prior to organ recovery.
10. Known hypersensitivity to human monoclonal antibodies or any of the study drug excipients.
11. Previous hypersensitivity to basiliximab, Campath-1H or antithymocyte globulin (ATG).
12. History of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin, or cervical intraepithelial neoplasia.
13. HIV positive recipients.
14. Hepatitis B surface antigen positive kidney transplant recipients.
15. Hepatitis B core antibody positive kidney transplant recipients.
16. Hepatitis C virus positive (HCV+) patients who are either untreated or have failed to demonstrate sustained viral remission for more than 12 months after anti-viral treatment.
17. Presence of clinically significant infections requiring continued therapy.
18. Positive screening for active tuberculosis.
19. Existence of any surgical or medical condition, other than the current transplantation which, in the opinion of the investigator, might significantly alter the distribution, metabolism or excretion of study medication.
20. Has a positive T- or B-cell cross-match by NIH anti-globulin lymphocytotoxicity method or CDC crossmatch method, if performed.
21. Has a positive T- or B-cell flow cross-match (over 250 channel shift) AND donor specific anti-HLA antibody (DSA) detected by flow cytometry (Luminex®) based antigen-specific anti-HLA antibody testing (over 4000 MFI) or by similar methodology, if performed.
22. History or presence of a medical condition or disease that in the investigator's assessment would place the patient at an unacceptable risk for study participation.
23. Lactating or pregnant woman.
24. Patient institutionalized by administrative or court order.
25. HLA or ABO incompatible kidney defined as a positive cytotoxic crossmatch or positive flow cross match.
26. Patients with known prothrombotic disorder (e.g. homozygous factor V leiden)
27. History of thrombosis or hypercoagulable state excluding access clotting
28. History of administration of C1INH containing products or recombinant C1INH within 15 days prior to study entry.
29. Patient with an abnormal Thromboelastogram.- results must be reported out prior to dosing (Defined by Coagulation Index of >3.0)
30. Patients on warfarin or other anti-coagulants or anti-platelets, such as Plavix, low molecular weight heparin (Low-dose aspirin prophylaxis allowed) due to a history or thrombotic or embolic events, or at a significantly increased risk for thrombosis due to conditions such as carotid stenosis or prosthetic valves.
31. Patients with known contraindication to treatment with C1INH
32. Patients with elevated abnormal platelet function (PLT>500,000).
33. Known or suspected allergy to rabbits and rabbit-derived products. History of immediate hypersensitivity reactions, including anaphylaxis, to C1 esterase inhibitor preparations.
34. Patients belonging to vulnerable populations: refers to but not limited to children, minors, pregnant women, prisoners, terminally ill patients, comatose, physically and intellectually challenged individuals, institutionalized, visual or hearing impaired, refugees, international research, and educationally disabled healthy volunteers.
35. Diagnosis of reversible Acute Kidney Injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-21 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients that do not meet DGF criteria based on creatinine levels following kidney transplantation from DCD donor who are treated with study drug compared to placebo | over a 12 month period
  Incidence of delayed graft function in the first 7 days following kidney transplant as defined as the initiation of dialysis in the first 7-days post transplantation and functional DGF as defined as a failure of the serum creatinine to decrease by at least 10% daily on 3 successive days during the first week post transplantation.

SECONDARY OUTCOMES:
Incidence of adverse and serious adverse events will be assessed via descriptive statistics method | over a 12 month period
  The feasibility of different statistical methods to analyze the incidence of adverse and serious adverse events
Ascertain whether any unexpected toxicities will occur in this patient population according to the Common Toxicity Criteria for Adverse Events (CTCAE) patient population | over a 12 month period
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Willingness of participation will be evaluated based on number of potential study candidates (approaches) compared to the number of candidates that enroll in the study likely response rates | over a 12 month period
  Enrollment rate of eligible participants
Tolerability following drug administration as measured by blood pressure | over a 12 month period
  The ability and tolerability to administer the study drug 3 times with appropriate post administration by recording blood pressure in mmHg
Tolerability following drug administration as measured by HR (heart rate) | over a 12 month period
  The ability and tolerability to administer the study drug 3 times with appropriate pre and post administration by recording heart rate as beats per minute
Tolerability following drug administration as measured by temperature | over a 12 month period
  The ability and tolerability to administer the study drug 3 times with appropriate pre and post administration by recording temperature in degrees Fahrenheit
Tolerability following drug administration as measured by respiratory rate | over a 12 month period
  The ability and tolerability to administer the study drug 3 times with appropriate pre and post administration by recording the respiratory rate as breathes per minute
Tolerability of drug administration as measured by urinary output | over a 12 month period
  To assess tolerability, upon administration of the drug, amount of urinary output will be recorded in mL

CONTACTS AND LOCATIONS:
Overall Officials: Luis Fernandez, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ricklin D, Hajishengallis G, Yang K, Lambris JD. Complement: a key system for immune surveillance and homeostasis. Nat Immunol. 2010 Sep;11(9):785-97. doi: 10.1038/ni.1923. Epub 2010 Aug 19. PMID 20720586
- [Background] Ricklin D, Lambris JD. Complement in immune and inflammatory disorders: pathophysiological mechanisms. J Immunol. 2013 Apr 15;190(8):3831-8. doi: 10.4049/jimmunol.1203487. PMID 23564577
- [Background] Zipfel PF, Skerka C. Complement regulators and inhibitory proteins. Nat Rev Immunol. 2009 Oct;9(10):729-40. doi: 10.1038/nri2620. Epub 2009 Sep 4. PMID 19730437
- [Background] Blom AM, Villoutreix BO, Dahlback B. Complement inhibitor C4b-binding protein-friend or foe in the innate immune system? Mol Immunol. 2004 Apr;40(18):1333-46. doi: 10.1016/j.molimm.2003.12.002. PMID 15072852
- [Background] Jozsi M, Zipfel PF. Factor H family proteins and human diseases. Trends Immunol. 2008 Aug;29(8):380-7. doi: 10.1016/j.it.2008.04.008. Epub 2008 Jul 2. PMID 18602340
- [Background] Davis AE 3rd. Biological effects of C1 inhibitor. Drug News Perspect. 2004 Sep;17(7):439-46. doi: 10.1358/dnp.2004.17.7.863703. PMID 15514703
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Kono H, Rock KL. How dying cells alert the immune system to danger. Nat Rev Immunol. 2008 Apr;8(4):279-89. doi: 10.1038/nri2215. Epub 2008 Mar 14. PMID 18340345
- [Background] Friedewald JJ, Rabb H. Inflammatory cells in ischemic acute renal failure. Kidney Int. 2004 Aug;66(2):486-91. doi: 10.1111/j.1523-1755.2004.761_3.x. PMID 15253694
- [Background] Diepenhorst GM, van Gulik TM, Hack CE. Complement-mediated ischemia-reperfusion injury: lessons learned from animal and clinical studies. Ann Surg. 2009 Jun;249(6):889-99. doi: 10.1097/SLA.0b013e3181a38f45. PMID 19474697
- [Background] Guo RF, Ward PA. Role of C5a in inflammatory responses. Annu Rev Immunol. 2005;23:821-52. doi: 10.1146/annurev.immunol.23.021704.115835. PMID 15771587
- [Background] McCaughan JA, O'Rourke DM, Courtney AE. The complement cascade in kidney disease: from sideline to center stage. Am J Kidney Dis. 2013 Sep;62(3):604-14. doi: 10.1053/j.ajkd.2012.12.033. Epub 2013 Mar 13. PMID 23489674
- [Background] Gasque P. Complement: a unique innate immune sensor for danger signals. Mol Immunol. 2004 Nov;41(11):1089-98. doi: 10.1016/j.molimm.2004.06.011. PMID 15476920
- [Background] Zhou W, Farrar CA, Abe K, Pratt JR, Marsh JE, Wang Y, Stahl GL, Sacks SH. Predominant role for C5b-9 in renal ischemia/reperfusion injury. J Clin Invest. 2000 May;105(10):1363-71. doi: 10.1172/JCI8621. PMID 10811844
- [Background] Weiser MR, Williams JP, Moore FD Jr, Kobzik L, Ma M, Hechtman HB, Carroll MC. Reperfusion injury of ischemic skeletal muscle is mediated by natural antibody and complement. J Exp Med. 1996 May 1;183(5):2343-8. doi: 10.1084/jem.183.5.2343. PMID 8642343
- [Background] de Vries B, Walter SJ, Peutz-Kootstra CJ, Wolfs TG, van Heurn LW, Buurman WA. The mannose-binding lectin-pathway is involved in complement activation in the course of renal ischemia-reperfusion injury. Am J Pathol. 2004 Nov;165(5):1677-88. doi: 10.1016/S0002-9440(10)63424-4. PMID 15509537
- [Background] Moller-Kristensen M, Wang W, Ruseva M, Thiel S, Nielsen S, Takahashi K, Shi L, Ezekowitz A, Jensenius JC, Gadjeva M. Mannan-binding lectin recognizes structures on ischaemic reperfused mouse kidneys and is implicated in tissue injury. Scand J Immunol. 2005 May;61(5):426-34. doi: 10.1111/j.1365-3083.2005.01591.x. PMID 15882434
- [Background] Schwaeble WJ, Lynch NJ, Clark JE, Marber M, Samani NJ, Ali YM, Dudler T, Parent B, Lhotta K, Wallis R, Farrar CA, Sacks S, Lee H, Zhang M, Iwaki D, Takahashi M, Fujita T, Tedford CE, Stover CM. Targeting of mannan-binding lectin-associated serine protease-2 confers protection from myocardial and gastrointestinal ischemia/reperfusion injury. Proc Natl Acad Sci U S A. 2011 May 3;108(18):7523-8. doi: 10.1073/pnas.1101748108. Epub 2011 Apr 18. PMID 21502512
- [Background] Castellano G, Melchiorre R, Loverre A, Ditonno P, Montinaro V, Rossini M, Divella C, Battaglia M, Lucarelli G, Annunziata G, Palazzo S, Selvaggi FP, Staffieri F, Crovace A, Daha MR, Mannesse M, van Wetering S, Paolo Schena F, Grandaliano G. Therapeutic targeting of classical and lectin pathways of complement protects from ischemia-reperfusion-induced renal damage. Am J Pathol. 2010 Apr;176(4):1648-59. doi: 10.2353/ajpath.2010.090276. Epub 2010 Feb 11. PMID 20150432
- [Background] Berger SP, Roos A, Mallat MJ, Fujita T, de Fijter JW, Daha MR. Association between mannose-binding lectin levels and graft survival in kidney transplantation. Am J Transplant. 2005 Jun;5(6):1361-6. doi: 10.1111/j.1600-6143.2005.00841.x. PMID 15888042
- [Background] Straatsburg IH, Boermeester MA, Wolbink GJ, van Gulik TM, Gouma DJ, Frederiks WM, Hack CE. Complement activation induced by ischemia-reperfusion in humans: a study in patients undergoing partial hepatectomy. J Hepatol. 2000 May;32(5):783-91. doi: 10.1016/s0168-8278(00)80247-0. PMID 10845665
- [Background] Williams JP, Pechet TT, Weiser MR, Reid R, Kobzik L, Moore FD Jr, Carroll MC, Hechtman HB. Intestinal reperfusion injury is mediated by IgM and complement. J Appl Physiol (1985). 1999 Mar;86(3):938-42. doi: 10.1152/jappl.1999.86.3.938. PMID 10066708
- [Background] Jordan JE, Montalto MC, Stahl GL. Inhibition of mannose-binding lectin reduces postischemic myocardial reperfusion injury. Circulation. 2001 Sep 18;104(12):1413-8. doi: 10.1161/hc3601.095578. PMID 11560858
- [Background] Sacks SH. Complement fragments C3a and C5a: the salt and pepper of the immune response. Eur J Immunol. 2010 Mar;40(3):668-70. doi: 10.1002/eji.201040355. PMID 20186746
- [Background] Peng Q, Li K, Smyth LA, Xing G, Wang N, Meader L, Lu B, Sacks SH, Zhou W. C3a and C5a promote renal ischemia-reperfusion injury. J Am Soc Nephrol. 2012 Sep;23(9):1474-85. doi: 10.1681/ASN.2011111072. Epub 2012 Jul 12. PMID 22797180
- [Background] de Vries B, Kohl J, Leclercq WK, Wolfs TG, van Bijnen AA, Heeringa P, Buurman WA. Complement factor C5a mediates renal ischemia-reperfusion injury independent from neutrophils. J Immunol. 2003 Apr 1;170(7):3883-9. doi: 10.4049/jimmunol.170.7.3883. PMID 12646657
- [Background] Djamali A, Muth BL, Ellis TM, Mohamed M, Fernandez LA, Miller KM, Bellingham JM, Odorico JS, Mezrich JD, Pirsch JD, D'Alessandro TM, Vidyasagar V, Hofmann RM, Torrealba JR, Kaufman DB, Foley DP. Increased C4d in post-reperfusion biopsies and increased donor specific antibodies at one-week post transplant are risk factors for acute rejection in mild to moderately sensitized kidney transplant recipients. Kidney Int. 2013 Jun;83(6):1185-92. doi: 10.1038/ki.2013.44. Epub 2013 Feb 27. PMID 23447068
- [Background] Stegall MD, Diwan T, Raghavaiah S, Cornell LD, Burns J, Dean PG, Cosio FG, Gandhi MJ, Kremers W, Gloor JM. Terminal complement inhibition decreases antibody-mediated rejection in sensitized renal transplant recipients. Am J Transplant. 2011 Nov;11(11):2405-13. doi: 10.1111/j.1600-6143.2011.03757.x. Epub 2011 Sep 22. PMID 21942930
- [Background] Lefaucheur C, Loupy A, Hill GS, Andrade J, Nochy D, Antoine C, Gautreau C, Charron D, Glotz D, Suberbielle-Boissel C. Preexisting donor-specific HLA antibodies predict outcome in kidney transplantation. J Am Soc Nephrol. 2010 Aug;21(8):1398-406. doi: 10.1681/ASN.2009101065. Epub 2010 Jul 15. PMID 20634297
- [Background] Lerut E, Naesens M, Kuypers DR, Vanrenterghem Y, Van Damme B. Subclinical peritubular capillaritis at 3 months is associated with chronic rejection at 1 year. Transplantation. 2007 Jun 15;83(11):1416-22. doi: 10.1097/01.tp.0000266676.10550.70. PMID 17565313
- [Background] Dean PG, Park WD, Cornell LD, Gloor JM, Stegall MD. Intragraft gene expression in positive crossmatch kidney allografts: ongoing inflammation mediates chronic antibody-mediated injury. Am J Transplant. 2012 Jun;12(6):1551-63. doi: 10.1111/j.1600-6143.2011.03964.x. Epub 2012 Feb 15. PMID 22335458
- [Background] Andres A, Marcen R, Valdes F, Plumed JS, Sola R, Errasti P, Lauzurica R, Pallardo L, Bustamante J, Amenabar JJ, Plaza JJ, Gomez E, Grinyo JM, Rengel M, Puig JM, Sanz A, Asensio C, Andres I; NI2A Study Group. A randomized trial of basiliximab with three different patterns of cyclosporin A initiation in renal transplant from expanded criteria donors and at high risk of delayed graft function. Clin Transplant. 2009 Jan-Feb;23(1):23-32. doi: 10.1111/j.1399-0012.2008.00891.x. Epub 2008 Sep 16. PMID 18798851
- [Background] Reddy KS, Stratta RJ, Alloway RR, Lo A, Hodge EE; PIVOT Study Group. The impact of delayed graft function of the kidney on the pancreas allograft in simultaneous kidney-pancreas transplantation. Transplant Proc. 2004 May;36(4):1078-9. doi: 10.1016/j.transproceed.2004.04.052. PMID 15194374
- [Background] Shoskes DA, Cecka JM. Effect of delayed graft function on short- and long-term kidney graft survival. Clin Transpl. 1997:297-303. PMID 9919413
- [Background] Sanfilippo F, Vaughn WK, Spees EK, Lucas BA. The detrimental effects of delayed graft function in cadaver donor renal transplantation. Transplantation. 1984 Dec;38(6):643-8. doi: 10.1097/00007890-198412000-00019. PMID 6390827
- [Background] Shoskes DA, Cecka JM. Deleterious effects of delayed graft function in cadaveric renal transplant recipients independent of acute rejection. Transplantation. 1998 Dec 27;66(12):1697-701. doi: 10.1097/00007890-199812270-00022. PMID 9884262
- [Background] Yokoyama I, Uchida K, Kobayashi T, Tominaga Y, Orihara A, Takagi H. Effect of prolonged delayed graft function on long-term graft outcome in cadaveric kidney transplantation. Clin Transplant. 1994 Apr;8(2 Pt 1):101-6. PMID 8019017
- [Background] Rosenthal JT, Danovitch GM, Wilkinson A, Ettenger RB. The high cost of delayed graft function in cadaveric renal transplantation. Transplantation. 1991 May;51(5):1115-8. No abstract available. PMID 2031264
- [Background] Matas AJ, Gillingham KJ, Elick BA, Dunn DL, Gruessner RW, Payne WD, Sutherland DE, Najarian JS. Risk factors for prolonged hospitalization after kidney transplants. Clin Transplant. 1997 Aug;11(4):259-64. PMID 9267712
- [Background] Floerchinger B, Oberhuber R, Tullius SG. Effects of brain death on organ quality and transplant outcome. Transplant Rev (Orlando). 2012 Apr;26(2):54-9. doi: 10.1016/j.trre.2011.10.001. PMID 22459036
- [Background] Danobeitia JS, Sperger JM, Hanson MS, Park EE, Chlebeck PJ, Roenneburg DA, Sears ML, Connor JX, Schwarznau A, Fernandez LA. Early activation of the inflammatory response in the liver of brain-dead non-human primates. J Surg Res. 2012 Aug;176(2):639-48. doi: 10.1016/j.jss.2011.10.042. Epub 2011 Nov 19. PMID 22440934
- [Background] van der Hoeven JA, Molema G, Ter Horst GJ, Freund RL, Wiersema J, van Schilfgaarde R, Leuvenink HG, Ploeg RJ. Relationship between duration of brain death and hemodynamic (in)stability on progressive dysfunction and increased immunologic activation of donor kidneys. Kidney Int. 2003 Nov;64(5):1874-82. doi: 10.1046/j.1523-1755.2003.00272.x. PMID 14531823
- [Background] Damman J, Schuurs TA, Ploeg RJ, Seelen MA. Complement and renal transplantation: from donor to recipient. Transplantation. 2008 Apr 15;85(7):923-7. doi: 10.1097/TP.0b013e3181683cf5. PMID 18408568
- [Background] Pratt JR, Abe K, Miyazaki M, Zhou W, Sacks SH. In situ localization of C3 synthesis in experimental acute renal allograft rejection. Am J Pathol. 2000 Sep;157(3):825-31. doi: 10.1016/S0002-9440(10)64596-8. PMID 10980122
- [Background] Damman J, Nijboer WN, Schuurs TA, Leuvenink HG, Morariu AM, Tullius SG, van Goor H, Ploeg RJ, Seelen MA. Local renal complement C3 induction by donor brain death is associated with reduced renal allograft function after transplantation. Nephrol Dial Transplant. 2011 Jul;26(7):2345-54. doi: 10.1093/ndt/gfq717. Epub 2010 Dec 2. PMID 21127132
- [Background] Atkinson C, Varela JC, Tomlinson S. Complement-dependent inflammation and injury in a murine model of brain dead donor hearts. Circ Res. 2009 Nov 20;105(11):1094-101. doi: 10.1161/CIRCRESAHA.109.194977. Epub 2009 Oct 8. PMID 19815824
- [Background] Damman J, Hoeger S, Boneschansker L, Theruvath A, Waldherr R, Leuvenink HG, Ploeg RJ, Yard BA, Seelen MA. Targeting complement activation in brain-dead donors improves renal function after transplantation. Transpl Immunol. 2011 May;24(4):233-7. doi: 10.1016/j.trim.2011.03.001. Epub 2011 Apr 1. PMID 21440065
- [Background] Naesens M, Li L, Ying L, Sansanwal P, Sigdel TK, Hsieh SC, Kambham N, Lerut E, Salvatierra O, Butte AJ, Sarwal MM. Expression of complement components differs between kidney allografts from living and deceased donors. J Am Soc Nephrol. 2009 Aug;20(8):1839-51. doi: 10.1681/ASN.2008111145. Epub 2009 May 14. PMID 19443638
- [Background] van Werkhoven MB, Damman J, van Dijk MCRF, Daha MR, de Jong IJ, Leliveld A, Krikke C, Leuvenink HG, van Goor H, van Son WJ, Olinga P, Hillebrands JL, Seelen MAJ. Complement mediated renal inflammation induced by donor brain death: role of renal C5a-C5aR interaction. Am J Transplant. 2013 Apr;13(4):875-882. doi: 10.1111/ajt.12130. Epub 2013 Feb 7. PMID 23398742
- [Background] Blogowski W, Dolegowska B, Salata D, Budkowska M, Domanski L, Starzynska T. Clinical analysis of perioperative complement activity during ischemia/reperfusion injury following renal transplantation. Clin J Am Soc Nephrol. 2012 Nov;7(11):1843-51. doi: 10.2215/CJN.02200312. Epub 2012 Aug 16. PMID 22904122
- [Background] de Vries DK, van der Pol P, van Anken GE, van Gijlswijk DJ, Damman J, Lindeman JH, Reinders ME, Schaapherder AF, Kooten Cv. Acute but transient release of terminal complement complex after reperfusion in clinical kidney transplantation. Transplantation. 2013 Mar 27;95(6):816-20. doi: 10.1097/TP.0b013e31827e31c9. PMID 23348894
- [Background] Davis AE 3rd, Lu F, Mejia P. C1 inhibitor, a multi-functional serine protease inhibitor. Thromb Haemost. 2010 Nov;104(5):886-93. doi: 10.1160/TH10-01-0073. Epub 2010 Aug 30. PMID 20806108
- [Background] Frank MM. Recombinant and plasma-purified human c1 inhibitor for the treatment of hereditary angioedema. World Allergy Organ J. 2010 Sep;3(9 Suppl):S29-33. doi: 10.1097/WOX.0b013e3181f1428d. PMID 23282867
- [Background] Curci C, Castellano G, Stasi A, Divella C, Loverre A, Gigante M, Simone S, Cariello M, Montinaro V, Lucarelli G, Ditonno P, Battaglia M, Crovace A, Staffieri F, Oortwijn B, van Amersfoort E, Gesualdo L, Grandaliano G. Endothelial-to-mesenchymal transition and renal fibrosis in ischaemia/reperfusion injury are mediated by complement anaphylatoxins and Akt pathway. Nephrol Dial Transplant. 2014 Apr;29(4):799-808. doi: 10.1093/ndt/gft516. Epub 2014 Jan 23. PMID 24463188
- [Background] Tillou X, Poirier N, Le Bas-Bernardet S, Hervouet J, Minault D, Renaudin K, Vistoli F, Karam G, Daha M, Soulillou JP, Blancho G. Recombinant human C1-inhibitor prevents acute antibody-mediated rejection in alloimmunized baboons. Kidney Int. 2010 Jul;78(2):152-9. doi: 10.1038/ki.2010.75. Epub 2010 Mar 24. PMID 20336054
- [Background] Sommer W, Tudorache I, Kuhn C, Avsar M, Salman J, Ius F, Gras C, Weber P, Welte T, Gottlieb J, Haverich A, Warnecke G. C1-esterase-inhibitor for primary graft dysfunction in lung transplantation. Transplantation. 2014 Jun 15;97(11):1185-91. doi: 10.1097/TP.0000000000000034. PMID 24573112
- [Background] Feldman HI, Gayner R, Berlin JA, Roth DA, Silibovsky R, Kushner S, Brayman KL, Burns JE, Kobrin SM, Friedman AL, Grossman RA. Delayed function reduces renal allograft survival independent of acute rejection. Nephrol Dial Transplant. 1996 Jul;11(7):1306-13. PMID 8672027
- [Background] Westendorp WH, Leuvenink HG, Ploeg RJ. Brain death induced renal injury. Curr Opin Organ Transplant. 2011 Apr;16(2):151-6. doi: 10.1097/MOT.0b013e328344a5dc. PMID 21415817
- [Background] Kim IK, Bedi DS, Denecke C, Ge X, Tullius SG. Impact of innate and adaptive immunity on rejection and tolerance. Transplantation. 2008 Oct 15;86(7):889-94. doi: 10.1097/TP.0b013e318186ac4a. PMID 18852649
- [Background] Damman J, Daha MR, van Son WJ, Leuvenink HG, Ploeg RJ, Seelen MA. Crosstalk between complement and Toll-like receptor activation in relation to donor brain death and renal ischemia-reperfusion injury. Am J Transplant. 2011 Apr;11(4):660-9. doi: 10.1111/j.1600-6143.2011.03475.x. PMID 21446970
- [Background] Asgari E, Zhou W, Sacks S. Complement in organ transplantation. Curr Opin Organ Transplant. 2010 Aug;15(4):486-91. doi: 10.1097/MOT.0b013e32833b9cb7. PMID 20631616
- [Background] Rao PS, Schaubel DE, Guidinger MK, Andreoni KA, Wolfe RA, Merion RM, Port FK, Sung RS. A comprehensive risk quantification score for deceased donor kidneys: the kidney donor risk index. Transplantation. 2009 Jul 27;88(2):231-6. doi: 10.1097/TP.0b013e3181ac620b. PMID 19623019
- [Background] Merion RM, Ashby VB, Wolfe RA, Distant DA, Hulbert-Shearon TE, Metzger RA, Ojo AO, Port FK. Deceased-donor characteristics and the survival benefit of kidney transplantation. JAMA. 2005 Dec 7;294(21):2726-33. doi: 10.1001/jama.294.21.2726. PMID 16333008
- [Background] Solez K, Colvin RB, Racusen LC, Haas M, Sis B, Mengel M, Halloran PF, Baldwin W, Banfi G, Collins AB, Cosio F, David DS, Drachenberg C, Einecke G, Fogo AB, Gibson IW, Glotz D, Iskandar SS, Kraus E, Lerut E, Mannon RB, Mihatsch M, Nankivell BJ, Nickeleit V, Papadimitriou JC, Randhawa P, Regele H, Renaudin K, Roberts I, Seron D, Smith RN, Valente M. Banff 07 classification of renal allograft pathology: updates and future directions. Am J Transplant. 2008 Apr;8(4):753-60. doi: 10.1111/j.1600-6143.2008.02159.x. Epub 2008 Feb 19. PMID 18294345
- [Background] Kaminska D, Koscielska-Kasprzak K, Drulis-Fajdasz D, Halon A, Polak W, Chudoba P, Janczak D, Mazanowska O, Patrzalek D, Klinger M. Kidney ischemic injury genes expressed after donor brain death are predictive for the outcome of kidney transplantation. Transplant Proc. 2011 Oct;43(8):2891-4. doi: 10.1016/j.transproceed.2011.08.062. PMID 21996181
- [Background] Parikh CR, Jani A, Mishra J, Ma Q, Kelly C, Barasch J, Edelstein CL, Devarajan P. Urine NGAL and IL-18 are predictive biomarkers for delayed graft function following kidney transplantation. Am J Transplant. 2006 Jul;6(7):1639-45. doi: 10.1111/j.1600-6143.2006.01352.x. PMID 16827865
- [Background] Waikar SS, Liu KD, Chertow GM. Diagnosis, epidemiology and outcomes of acute kidney injury. Clin J Am Soc Nephrol. 2008 May;3(3):844-61. doi: 10.2215/CJN.05191107. Epub 2008 Mar 12. PMID 18337550
- [Background] Damman J, Kok JL, Snieder H, Leuvenink HG, van Goor H, Hillebrands JL, van Dijk MC, Hepkema BG, Reznichenko A, van den Born J, de Borst MH, Bakker SJ, Navis GJ, Ploeg RJ, Seelen MA. Lectin complement pathway gene profile of the donor and recipient does not influence graft outcome after kidney transplantation. Mol Immunol. 2012 Feb;50(1-2):1-8. doi: 10.1016/j.molimm.2011.11.009. Epub 2011 Dec 15. PMID 22173059
- [Background] Heijnen BH, Straatsburg IH, Padilla ND, Van Mierlo GJ, Hack CE, Van Gulik TM. Inhibition of classical complement activation attenuates liver ischaemia and reperfusion injury in a rat model. Clin Exp Immunol. 2006 Jan;143(1):15-23. doi: 10.1111/j.1365-2249.2005.02958.x. PMID 16367929